CLINICAL TRIAL: NCT04994314
Title: Effect of Calcium Fluoride Nanoparticles in Prevention of Demineralization During Orthodontic Fixed Appliance Treatment: a Randomized Clinical Trial
Brief Title: White Spot Lesions Prevention During Orthodontic Fixed Appliance Treatment: a Randomized Clinical Trial
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Baghdad (Other)
Responsible Party: Principal Investigator, Rawof Rasheed Jawad, Assistant professor, University of Baghdad
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: calcium fluoride nanoparticles
Record Dates: First submitted 2021-07-27; First posted 2021-08-06 (Actual); Last update posted 2021-08-06 (Actual); Status verified 2021-08

CONDITIONS: White Spot Lesion of Tooth
Keywords: white spot lesions; orthodontic primer; calcium fluoride nanoparticles

STUDY DESIGN:
Intervention Model Description: The study planned to be split mouth study with equal randomization (1:1 allocation ratio)
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This study proposed to be double blinded (the patients, investigators and the outcome assessors)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- orthodontic primer containing calcium fluoride nanoparticles (Active Comparator): Fixed appliance for ten maxillary teeth and the contralateral mandibular teeth will be bonded using orthodontic primer containing calcium fluoride nanoparticles
  Interventions: Drug: nCaF2 primer
- Control primer (Placebo Comparator): Fixed appliance for ten maxillary teeth (contralateral to experimental ten side)and the contralateral mandibular teeth will be bonded using conventional primer (TransbondTM XT orthodontic primers (3M-Unitek, Monrovia, USA)
  Interventions: Drug: Control primer

INTERVENTIONS:
Drug: nCaF2 primer — Calcium fluoride nanoparticles was added to conventional orthodontic primers to develop bioactive primer. This primer was examined previously for its biological and physical properties
  Other Names: Orthodontic primer containing calcium fluoride nanoparticles
  Arms: orthodontic primer containing calcium fluoride nanoparticles
Drug: Control primer — Conventional orthodontic primer
  Other Names: TransbondTM XT orthodontic primer
  Arms: Control primer

SUMMARY:
The aim of this study is to evaluate the effectiveness of calcium fluoride nanoparticles containing orthodontic primer in preventing or decreasing the incidence WSLs over a period of 6 months in patients with fixed orthodontic appliances.

This study proposed to be double blinded, split mouth, randomized clinical trial, with equal randomization (1:1 allocation ratio).

DETAILED DESCRIPTION:
The sample was selected and recruited from patients attending two centres (Orthodontic Department at Karbala Governmental Specialized Dental Center and Almina Dental Private Clinics/Karbala), but the bonding and follow up sessions were done in Almina Dental Private Clinics/Karbala. Patient recruitment was done according to specified inclusion and exclusion criteria.

Intervention procedure planned to be by bonding fixed orthodontic appliances to all patients. The four quadrants of the mouth will be divided into two groups (Group 1 and 2), with one group, the upper right and lower left quadrants bonded with nCaF2 resin, while the upper left and lower right quadrants bonded with control resin. For the other group, the reverse will be carried out. Then, by the use of a computer random number generator, the two groups will be randomly allocated, and each number in the random table will be given a study number in order to create the final Allocation Table for the participants in the study (which contained the study number and allocation group). the primary planned to be measured by DIAGNOdent Pen 2190 device to measure enamel demineralization objectively, while the secondary objective planned to be quantitative detection of Streptococcus mutans bacteria by using real-time PCR

ELIGIBILITY:
Inclusion Criteria:

* Patients have

  1. Fully erupted permanent teeth (regardless the third molar),
  2. Indication to have orthodontic treatment without extraction
  3. Fair or good oral hygiene before or after oral hygiene instruction

Exclusion Criteria:

* Patients will be excluded if they had

  1. Previous orthodontic treatment or extractions
  2. Missing teeth
  3. Active enamel caries determined by clinical examination
  4. Patients with enamel hypoplasia, dental fluorosis or tetracycline pigmentation
  5. Labial restorations
  6. Severe periodontal diseases determined according to PDI index by Sigurd P. Ramfjord (Ramfjord, 1967)
  7. Craniofacial syndromes such as clefts
  8. Xerostomia determined from clinical history of the patient
  9. Severely rotated teeth (limiting the appearance of buccal surfaces)
  10. Heavy smokers determined by accounting the number of cigarettes per day and time to the first cigarette of the day (Heatherton et al., 1989) .

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 31 (Estimated)
Dates: Start 2021-02-15 (Actual); Primary Completion 2021-12-16 (Estimated); Study Completion 2022-02-15 (Estimated)

PRIMARY OUTCOMES:
DIAGNOdent Pen scores change | Six months
  assessing changes in the amount of enamel demineralization (DIAGNOdent Pen scores) between four time points:-
  1. baseline (before brackets bonding)
  2. after one month of brackets bonding
  3. after three months of brackets bonding
  4. after six months of brackets bonding

SECONDARY OUTCOMES:
Streptococcus mutans load change | Six months
  Quantitative detection of streptococcus mutans load changes (using real time PCR) between four time points:-
  1. baseline (before brackets bonding)
  2. after one month of brackets bonding
  3. after three months of brackets bonding
  4. after six months of brackets bonding

CONTACTS AND LOCATIONS:
Overall Officials: Yassir A. Yassir, PhD, Study Director — Baghdad University- College of Dentistry
Locations (1):
- Almina dental clinics, Karbala, Iraq

REFERENCES:
- [Derived] Al Tuma RR, Yassir YA. Effect of calcium fluoride nanoparticles in prevention of demineralization during orthodontic fixed appliance treatment: a randomized clinical trial. Eur J Orthod. 2023 Mar 31;45(2):122-132. doi: 10.1093/ejo/cjac055. PMID 36049047